CLINICAL TRIAL: NCT00732862
Title: Metabolic Adaptation to Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Steve Davis, Chairman of Medicine, University of Maryland, Baltimore, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#8842-NIDDM
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; intensive therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucose Clamp Technique

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Baseline clamp study before treatment phase.
  Interventions: Procedure: glucose clamp
- 2 (Active Comparator): Final clamp experiment after 6 months intensive therapy.
  Interventions: Procedure: glucose clamp

INTERVENTIONS:
Procedure: glucose clamp — Hyperinsulinemic Hypoglycemic clamp
  Arms: 1
Procedure: glucose clamp — Hyperinsulinemic Hypoglycemic clamp
  Arms: 2

SUMMARY:
Hypoglycemia or low blood sugar is a very serious complication that diabetics experience. This is of great concern because there is a lack of available information of how Non Insulin Dependent Diabetic Mellitus patients (NIDDM) defend themselves against a low blood sugar. This is particularly disturbing since NIDDM patients are likely to require intensive treatment, and as a result, the risks of severe hypoglycemia to the NIDDM patient increase. The current proposal aims to provide information on how NIDDM patients can defend themselves against hypoglycemia, thus decreasing their risks for this severe complication.

DETAILED DESCRIPTION:
There is very little data available on the neuroendocrine response to hypoglycemia in intensively treated (sulfonylurea or insulin) NIDDM patients. The data that are available on the neuroendocrine response to hypoglycemia in NIDDM patients were obtained under conditions following a single IV bolus of insulin or single SQ regular insulin injection. The neuroendocrine response following a large IV bolus of insulin differs greatly from the clinical paradigm of a slow progression into hypoglycemia. Therefore, clinically relevant data cannot be obtained from short experiments involving rapid changes in plasma glucose levels and insulinemia. Furthermore, a comparison between neuroendocrine responses to hypoglycemia in NIDDM and normal man is not available due to the fact that glycemia has never been equally controlled. In short, virtually nothing is known about the neuroendocrine response to hypoglycemia in these subjects. This is of great concern as following the positive outcome of the Kumamato study, large numbers of NIDDM subjects are going to receive intensive therapy with all its altendent risks of severe hypoglycemia. The Kumamato study was a trial in NIDDM patients to determine if intensive therapy reduces tissue complications of diabetes. Similar to the results of the Diabetes control and complications trial in IDDM patients the Kumamato study proved that intensive therapy in NIDDM patients also prevents diabetic tissue complications. Therefore, the goals of this study are 1) to define in greater detail how the body defends itself against hypoglycemia in NIDDM patients and 2) to determine if differing levels of insulin affect hypoglycemic counterregulation in NIDDM patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 30-65 years
* Male and female non-insulin-dependent diabetic patients, sulfonylurea and/or Metformin aged 30-65 years

Exclusion Criteria:

* Prior or current history of poor health
* Abnormal results following screening tests
* Pregnancy

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 1998-02; Primary Completion 2000-03 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
HbA1c | 6 months

SECONDARY OUTCOMES:
Catecholamines | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen N Davis, MD, Principal Investigator — Vanderbilt University